CLINICAL TRIAL: NCT03542617
Title: Effect of Preoperative Intravenous Dexamethasone on Postoperative Pain After Primary Total Hip Arthroplasty : A Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Preoperative Intravenous Dexamethasone on Postoperative Pain After Primary Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Nitchanant Kitcharanant, Effect of Preoperative Intravenous Dexamethasone on Postoperative Pain After Primary Total Hip Arthroplasty : A prospective, double-blind, randomized controlled trial, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORT-2559-03928
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Localized Primary Osteoarthritis of Both Hips (Diagnosis); Osteoarthritis, Hip
MeSH Terms: conditions — Disease; Osteoarthritis, Hip | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline Solution (Placebo Comparator): The control group receive sterile normal saline solution, as placebo, intravenous immediately prior to induction of spinal anesthesia .
  Interventions: Drug: Normal Saline Solution
- 10 mg Dexamethasone (Active Comparator): The steroid group will receive Dexamethasone 10 mg IV immediately prior to induction of spinal anesthesia
  Interventions: Drug: Dexamethasone
- 40 mg Dexamethasone (Active Comparator): The steroid group will receive Dexamethasone 40 mg IV immediately prior to induction of spinal anesthesia
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone
  Arms: 10 mg Dexamethasone; 40 mg Dexamethasone
Drug: Normal Saline Solution
  Arms: Normal Saline Solution

SUMMARY:
To compare the effects of preoperative intravenous Dexamethasone between 10 mg and 40 mg with placebo on Postoperative Pain After Primary Total Hip Arthroplasty

DETAILED DESCRIPTION:
It still unclear whether the effective dose preoperative intravenous dexamethasone on postoperative pain after Total Hip Arthroplasty. The research hypothesis is that the effect of 10 mg intravenous Dexamethasone in postoperative pain(5 metre walking at 24 hour) is not inferior to 40 mg intravenous Dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Undergoing Elective, Primary, unilateral Total Hip arthroplasty
* American Society of Anesthesiology (ASA) physical class 1-3
* BMI < 40 kg/m2

Exclusion Criteria:

* History of previous musculoskeletal injury on the same hip
* History of prior surgery on the same unilateral hip
* History of adverse effects from medication utilized in this study
* Contraindication to spinal anesthesia
* History of psychiatric disorders or cognitive impairment
* Contraindication to Corticosteroid
* Poorly controlled Diabetes mellitus
* History of ischemic heart disease or peripheral arterial disease or cerebrovascular disease
* Hepatic insufficiency (Child-Pugh score > 5)
* Renal insufficiency (Creatinine clearance < 30 mL/min)
* History of cataract or glaucoma or ocular hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scales for pain during five-metre walking (0-100) | at 24 hours postoperatively
  Each pain outcome will be assessed using a visual analogue scale of 0-100 mm, in which 0 indicates no pain and 100 indicates the worst pain;

SECONDARY OUTCOMES:
Visual analogue scales for pain during five-metre walking (0-100) | Postoperative at 48,72 hours.
  Each pain outcome will be assessed using a visual analogue scale of 0-100 mm, in which 0 indicates no pain and 100 indicates the worst pain;
Visual analogue scales for pain on 45 degree active hip flexion (0-100) | Postoperative at 24,48,72 hours.
  Each pain outcome will be assessed using a visual analogue scale of 0-100 mm, in which 0 indicates no pain and 100 indicates the worst pain;
Visual analogue scales for current pain at rest on supine position (0-100) | Postoperative at 6,24,48,72 hours.
  Each pain outcome will be assessed using a visual analogue scale of 0-100 mm, in which 0 indicates no pain and 100 indicates the worst pain;
Visual analogue scales for the maximal pain at rest over the last 24 hours and the minimal pain at rest over the last 24 hours (0-100) | Postoperative at 0-24,24-48,48-72 hours.
  Each pain outcome will be assessed using a visual analogue scale of 0-100 mm, in which 0 indicates no pain and 100 indicates the worst pain;
Visual analogue scales for nausea (0-100) | Postoperative at 6,24,48,72 hours
  This outcome will be assessed in a form of visual analogue scale of 0-100 mm, in which 0 indicates no nausea or vomiting and 100 indicates the worst nausea or vomiting
Opioid consumption (mg.) | Postoperative at 0-24,24-48,48-72 hours
  Opioid consumption (mg.)
Anti-emetic medicine consumption (mg.) | Postoperative at 0-24,24-48,48-72 hours
  Anti-emetic medicine consumption (mg.)
Wound complication | Postoperative at Discharge, 2 weeks, 6 weeks, 12 weeks.
  Wound complications (including periprosthetic joint infection and inadequate wound healing). Periprosthetic joint infection will be diagnosed using the criteria outlined by the Musculoskeletal Infection Society. Inadequate wound healing is defined as delayed wound healing or wound dehiscence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Chiang Mai University, Chiang Mai, Thailand